CLINICAL TRIAL: NCT01627028
Title: Thai Traditional Massage Increases Biochemical Marker of Bone Formation in Postmenopausal Women: a Randomized Crossover Trial
Brief Title: Thai Traditional Massage Increases Biochemical Marker of Bone Formation in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: ID 10-53-28
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Osteoporosis
Keywords: Thai traditional massage; Bone formation; Bone resorption
MeSH Terms: conditions — Osteoporosis; Bone Resorption | interventions — Medicine, Thai Traditional

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Thai traditional massage — two hours of Thai traditional massage twice a week for 4 weeks

SUMMARY:
To investigate the skeletal effect of Thai traditional massage by examining the changes in biochemical markers of bone turnover.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women

EXclusion Criteria:

* History of hyperthyroidism, thyrotoxicosis, diabetes, rheumatoid arthritis and cancer
* glucocorticoid or medication for osteoporosis
* Swelling joints

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sampling
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Saetung S, Chailurkit LO, Ongphiphadhanakul B. Thai traditional massage increases biochemical markers of bone formation in postmenopausal women: a randomized crossover trial. BMC Complement Altern Med. 2013 Mar 25;13:69. doi: 10.1186/1472-6882-13-69. PMID 23530566